CLINICAL TRIAL: NCT07249866
Title: Effect of Robotic Assisted Therapy on Hand Functions, Grip Strength and Proprioception in Children With Hemiplegia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Attia El Shemy, professor and chairman of department of physical therapy for pediatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005785
Record Dates: First submitted 2025-08-25; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy, Spastic
Keywords: robotic therapy; hand functions; hemiplegia; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic assisted therapy (Experimental): robotic hand assisted therapy using robotic gloves for 8 weeks 3seesions / week each session lasts 30 minutes including passive , active assisted, active resisted, mirroring and gaming mode
  Interventions: Device: Hand rehabilitation robotic gloves; Other: occupational therapy
- Traditional occupational therapy (Active Comparator): 3 sessions/ week for 8 weeks and each session lasts 30 minutes using scissors - Knocking peg board with hammer- Building towers with rings-- Cubes insertion into wide muzzle jars- Playing with clays and form small balls and rolls
  Interventions: Other: occupational therapy

INTERVENTIONS:
Device: Hand rehabilitation robotic gloves — robotic gloves assist in hand functions
  Arms: Robotic assisted therapy
Other: occupational therapy — designed traditional occupational therapy program

SUMMARY:
Statement of the problem:

Does robotic assisted therapy have an effect on hand functions, grip strength and proprioception in children with hemiplegic cerebral palsy?

Significance of the study:

New technologies allow and promote active involvement, leading directly to functional changes that are far beyond those obtained with conventional therapy. Many features of robotic therapy may contribute to enhanced recovery of upper limb motor function. These include task-specific practice, intensity of repetition, robotic assistance, enhanced sensory feedback, continual motivation (because every trial yields a degree of success, even if robot assistance is required).

The implementation of robotics with hemiplegic cerebral palsy focuses on functional motor performance by providing intensive repetitive training, sensorimotor integration and cognitive engagement through goal-directed tasks to address the underlying symptoms. Robotic technologies offer numerous potential advantages over conventional therapies, chief among these being the ability to provide high-intensity repetitive training. Robotic treatment is a novel approach that has demonstrated promise in enhancing motor function, enhancing the quality of life, and lessening the burden on caregivers.

DETAILED DESCRIPTION:
Thirty two children with hemiplegic cerebral palsy from both sexes according to G*power analysis (α= 0.05 , Power= 0.90 , effect size = 0.89) Their ages range from 6- 9 years. Mild to moderate degree of spasticity, according to modified Ashworth scale (grade 1 to 2).

Motor function level will be I and II according to gross motor function classification system.

Assessment will be conducted using Bruininks Oseretsky test of motor proficiency scale 2nd edition (BOT-2) for assessment of fine motor control , handheld dynamometer will be used for measuring hand grip strength and digital goniometer for measuring wrist joint sense of position.

Children in the study group will receive robotic assisted therapy.

Null Hypothesis:

There will be no effect of robotic assisted therapy on hand functions, grip strength and proprioception in children with hemiplegic cerebral palsy .

Basic assumptions:

All children will attend the treatment program regularly. All children will follow the same sequence of the treatment procedure. All children will be cooperative and following the instructions during evaluation and treatment procedures.

The results of the study will be helpful for physical therapists dealing with children with the same condition

Inclusion Criteria:

Their ages range from 6-9 years. They have mild to moderate spasticity (grade 1- 2) according to Modified Ashworth Scale Their motor function will be at level I and II according to Gross Motor Function Classification System GMFCS Their manual abilities will be at level II and Level III according to Manual Ability classification system as mentioned in a previous review They will be able to understand and follow instructions

Exclusion criteria:

Fixed deformity in any joints of the upper limb. Previous history of surgical intervention in the upper limb. Auditory, visual and cognitive problems. Botulinum Toxin injection in last 6 months

ELIGIBILITY:
Inclusion Criteria:

* Their ages range from 6-9 years
* They have mild to moderate spasticity (grade 1- 2) according to Modified Ashworth Scale
* Their motor function will be at level I and II according to Gross Motor Function Classification System GMFCS
* Their manual abilities will be at level II and Level III according to Manual Ability classification system
* They will be able to understand and follow instructions

Exclusion Criteria:

* Fixed deformity in any joints of the upper limb.
* Previous history of surgical intervention in the upper limb.
* Auditory, visual and cognitive problems.
* Botulinum Toxin injection in last 6 months.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
hand grip strength by hand held dynamometer | 8 weeks
  the hand grip strength will be measured by hand held dynamometer
hand functions ( fine motor precision and integration measured by Bruininks-Oseretsky Test of Motor Proficiency | 8 weeks
  hand functions will be measured by Bruininks-Oseretsky Test of Motor Proficiency
wrist joint proprioception by digital goniometer | 8 weeks
  wrist joint position sense will be measured by digital goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Samah Attia El shemy, professor doctor, Principal Investigator — Cairo university, Faculty of physical therapy
Locations (1):
- Cairo University, Cairo, State/Province, Egypt

IPD SHARING:
Plan to Share IPD: No
any participant data will be available on direct request from authors